CLINICAL TRIAL: NCT02723409
Title: Umbilicoplasty: A Randomized Controlled Trial of Techniques for Umbilical Reconstruction Following Abdominoplasty and Abdominally-based Free Tissue Transfer
Brief Title: Trial of Techniques for Umbilical Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-00480
Record Dates: First submitted 2016-03-08; First posted 2016-03-30 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Umbilicoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Round Procedure (Active Comparator): umbilicoplasty technique
  Interventions: Procedure: Round Procedure Umbilicoplasty
- "Scarless" round procedure (Active Comparator): umbilicoplasty technique
  Interventions: Procedure: Scarless" round procedure
- "Inverted U" procedure (Active Comparator): umbilicoplasty technique
  Interventions: Procedure: "Inverted U" Procedure
- "Inverted V" procedure (Active Comparator): umbilicoplasty technique
  Interventions: Procedure: "Inverted V"Procedure
- Y deepithelialized" procedure (Active Comparator): umbilicoplasty technique
  Interventions: Procedure: "Y deepithelialized" Procedure

INTERVENTIONS:
Procedure: Round Procedure Umbilicoplasty — Umbilicoplasty surgery (belly button reshaping) is performed using the "Round Procedure"
  Arms: Round Procedure
Procedure: Scarless" round procedure — Umbilicoplasty surgery (belly button reshaping) is performed using the "Scarless" round procedure
  Arms: "Scarless" round procedure
Procedure: "Inverted U" Procedure — Umbilicoplasty surgery (belly button reshaping) is performed using the "Inverted U" Procedure
  Arms: "Inverted U" procedure
Procedure: "Inverted V"Procedure — Umbilicoplasty surgery (belly button reshaping) is performed using the "Inverted V" Procedure
  Arms: "Inverted V" procedure
Procedure: "Y deepithelialized" Procedure — Umbilicoplasty surgery (belly button reshaping) is performed using the "Y deepithelialized" procedure
  Arms: Y deepithelialized" procedure

SUMMARY:
The primary objective of the study will be to determine which of five traditionally used umbilical reconstructive techniques offers superior aesthetic results. Additionally, secondary objectives of post-operative complications such as hypertrophic scar formation will also be measured.

DETAILED DESCRIPTION:
This is a five arm, prospective, randomized, trial. Patients undergoing abdominoplasty or abdominally-based free tissue transfer (TRAM/DIEP flaps) at NYU Medical Center will be randomly assigned to receive one of five conventionally used umbilicoplasty techniques during the course of their surgery:

1. Round procedure
2. "Scarless" round procedure
3. "Inverted u" procedure
4. "Inverted v" procedure, and
5. "Y deepithelialized" procedure

As there has not yet been a superiority or inferiority comparison of these five methods, no patient will be receiving substandard care by randomization to one of the five procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Female patients undergoing abdominoplasty or abdominally-based free tissue transfer (TRAM/DIEP flaps)

Exclusion Criteria:

* Patients with prior history of umbilicoplasty
* History of keloid formation
* Active smokers
* Body Mass Index (BMI) over 40

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Change in measurement of patient assessment post-operative and pre-operative, using a VAS survey results with a positive result indicating a favorable outcome | Baseline, 12 Weeks
Assessment of inter-rater reliability among physicians in the assessment of the aesthetic outcomes of umbilical reconstruction. | 12 Weeks
Comparison of aesthetic outcomes of umbilical reconstruction using five accepted techniques for umbilicoplasty following abdominoplasty or abdominally-based free tissue transfer (TRAM/DIEP flaps). | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: VIshal Thanik, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States